CLINICAL TRIAL: NCT02904148
Title: Measurement of the Analgesic Efficacy of Shoulder Mobilization in Hemiplegic Patients
Brief Title: Passive Mobilisation of Region of Shoulder Joints for Hemiplegic Patient
Acronym: ERIAMS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015/CHU/09
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-07

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shoulder mobilisation (Experimental): The shoulder mobilisation is performed daily by a physiotherapist for 45 days.
  Interventions: Procedure: Shoulder mobilisation

INTERVENTIONS:
Procedure: Shoulder mobilisation — early shoulder mobilisation

SUMMARY:
Hemiplegia is a high prevalence pathology with 1 per 1000 habitants in France. One of these complications is shoulder pain which affects about 35 to 70% of cases. The medical care of this complication is critical because it affects the patient's quality of life and also hinders participation in rehabilitation sessions slowing the recovery of independence in activities of daily living.

Literature confirmed the involvement of the scapula in the hemiplegic shoulder pain with his attitude pronounced lateral rotation. But no data to confirm that passive mobilization reduce shoulder pain.

Because no data available to permit us to determine the sample size we set-up this preliminary study to check if efficiency found in these preliminary data are consistent with an estimable real efficacy in a randomized trial feasible.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in Physical Medicine and Rehabilitation at Centre Hospitalier Universitaire Réunion (Site of Le Tampon)
* Having made a cerebrovascular accident between 30 and 3 days before inclusion
* with pain in the upper limb whose score with visual analogue scale is greater than or equal to 20 mm
* able to understand the question: "Do you have arm pain?"

Exclusion Criteria:

* with visual analogue scale score lower than 20 mm at the inclusion
* with aphasia of comprehension
* with medical contraindication for passive shoulder mobilisation (Shoulder fracture, dislocation,...)
* opposing to any mobilization
* with shoulder pathology previously known
* history of cerebrovascular accident prior 30 days before inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Pain evaluation with visual analogic scale | Change of pain evaluation between Day 0 and Day 45
  Proportion of patients reducing by at least 20 mm their score on the visual analogic scale (VAS) from baseline Day 45

CONTACTS AND LOCATIONS:
Overall Officials: Andre Muller, MD, Principal Investigator — CHU de La Réunion

IPD SHARING:
Plan to Share IPD: No